CLINICAL TRIAL: NCT02225613
Title: Comparison Between Two Rehabilitation Programs (Conventional and Aquatic) After Cruciate Ligament Injury in Sportsmen
Brief Title: Spa Rehabilitation After Cruciate Ligament Injury in Sportsmen
Acronym: Thermasport
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A00390-47
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Cruciate Ligament Injury; Balance Control
Keywords: Cruciate ligament injury; Balance control; Rehabilitation; Spa therapy; Sport

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual protocol (Active Comparator): 2 weeks conventional rehabilitation 3 weeks conventional rehabilitation
  Interventions: Other: Usual protocol
- Spa protocol (Active Comparator): 2 weeks conventional rehabilitation 3 weeks aquatic rehabilitation
  Interventions: Other: Spa protocol

INTERVENTIONS:
Other: Usual protocol
  Arms: Usual protocol
Other: Spa protocol
  Arms: Spa protocol

SUMMARY:
Knee cruciate ligament injury is a common injury (15 000 per year in France) which concerns young sportsmen. Consequences are limitation in physical and sporting activities and at work.

Main objective: to compare water and traditional rehabilitation after cruciate ligament injury reconstruction in terms of kinematics of recovery and of proprioceptive abilities development.

DETAILED DESCRIPTION:
Secondary objectives: to compare algo-functional and sport, social and job come back date between both groups.

Multicentric randomised trial comparing two therapy protocols in knee cruciate ligament injury.

After surgery, 2 weeks rehabilitation; 3 weeks conventional rehabilitation (group 1) or rehabilitation in water (group 2).

Data will be collected at inclusion (before surgery), 2 weeks, 1 month, 2 months and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults,
* 18-49 years,
* indication of knee anterior cruciate ligament reconstruction.

Exclusion Criteria:

* other recent lower limb sprain,
* history of neurological disease (stroke, central or peripheral degenerative disease),
* psychtrope or antihypertensive drugs,
* aquatic activities contra-indication (cutaneous).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Posturography composite score | up to 6 months
  Postural control during quiet stance will be evaluated without and with sensory conflict by a sensory organization test

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Nancy, Lorraine, France

REFERENCES:
- [Derived] Peultier-Celli L, Mainard D, Wein F, Paris N, Boisseau P, Ferry A, Gueguen R, Chary-Valckenaere I, Paysant J, Perrin P. Comparison of an Innovative Rehabilitation, Combining Reduced Conventional Rehabilitation with Balneotherapy, and a Conventional Rehabilitation after Anterior Cruciate Ligament Reconstruction in Athletes. Front Surg. 2017 Nov 7;4:61. doi: 10.3389/fsurg.2017.00061. eCollection 2017. PMID 29164130